CLINICAL TRIAL: NCT01800266
Title: Improving Practice in Community-based Settings: A Randomized Trial of Supervision Strategies
Brief Title: Randomized Controlled Trial of Supervision Strategies to Improve Clinician Fidelity to Trauma-focused CBT
Acronym: STEPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Principal Investigator, Shannon Dorsey, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: A64442; R01MH095749 (NIH)
Record Dates: First submitted 2013-02-22; First posted 2013-02-27 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Post Traumatic Stress; Overall Functioning; Clinician Fidelity; Supervision
Keywords: Supervision; Implementation; Community Based Mental Health Services; Trauma Focused Cognitive Behavioral Therapy; Skill Building and Behavioral Rehearsal; Symptom and Fidelity Monitoring; Children; Adolescents
MeSH Terms: conditions — Assessment of Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Symptom and Fidelity Monitoring (SFM) (Experimental): Half of the study clinicians will be randomized to this supervision condition of TF-CBT.
  Interventions: Behavioral: Supervision Practices of TF-CBT
- SFM + Behavioral Rehearsal (Experimental): Half of the study clinicians will be randomized to this supervision condition of TF-CBT.
  Interventions: Behavioral: Supervision Practices of TF-CBT

INTERVENTIONS:
Behavioral: Supervision Practices of TF-CBT — Supervisors will be trained in one of two supervision strategies: Symptom and Fidelity Monitoring (SFM) or Symptom and Fidelity Monitoring + Behavioral Rehearsal (SFM + BR)

SUMMARY:
The primary goal of this study is to examine the impact of varying supervision strategies on clinician fidelity and client outcomes in a community-based setting. Prior research has established that training approaches that do not include a period of intervention-specific supervision or consultation are ineffective and that implementation efforts that include only an initial period of supervision show an eventual attenuation of gains in knowledge and fidelity in practice. Ongoing supervision may be required for effective and sustained implementation of evidence-based practices (EBPs) in community-based settings. However, supervision is one of the least investigated aspects of training. "Gold standard" elements of supervision from efficacy trials include review of sessions, standardized procedures for monitoring client outcomes and model fidelity, and ongoing skill-building (e.g., behavioral rehearsal). The degree (e.g., frequency, intensity) to which these strategies are used in community-based settings is unknown.

There are a growing number of national and statewide efforts to increase the reach of EBPs through dissemination and implementation initiatives. There are 18 statewide initiatives to implement Trauma-focused Cognitive Behavioral Therapy (TF-CBT), an EBP for child trauma exposure and sequelae. Many of the community based TF-CBT implementation efforts, and those for other EBPs, include a specific focus on supervisors. However, the limited scientific literature provides very little guidance for these efforts. Aims of the current trial include 1) studying supervision with existing implementation supports; particularly presence of gold standard elements; 2) evaluating the effects of varying supervision strategies on fidelity and client outcomes; and 3) testing the mediating effect of treatment fidelity on the relationship between supervision type and client outcomes. We propose a two-phased, within-subjects and between subjects design. In Phase I (9 months), we examined supervision with implementation support. In Phase II (30 months), we will examine two specific supervision conditions, each including varying EBP supervision elements.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6-17 who are starting Trauma-focused Cognitive Behavioral Therapy (TF-CBT) with one of our enrolled clinicians.They must also have significant Post Traumatic Stress symptoms as measured by a score of 21 or higher on the UCLA PTSD-RI, and live with a parent or guardian who is willing to participate in the study.
* Community-based mental health clinicians who are employed in Regional Support Network agencies (state Medicaid clinics) who have participated in the Washington State Initiative for TF-CBT and are supervised by a participating supervisor, or have completed the TF-CBT web training and been supervised on a case.
* Community-based mental health supervisors trained in the WA State Initiative in TF-CBT and employed at participating clinics in WA.

Exclusion Criteria:

* Non-English speaking child.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1280 (Estimated)
Dates: Start 2012-07; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Coding Therapy Sessions to Assess Clinician Fidelity to TF-CBT Strategy. | 2 years
  Evidence-Based Practices such as Trauma-focused Cognitive Behavioral Therapy (TF-CBT) usually include ongoing supervision to assess how true (e.g. fidelity) clinicians stay to their training in the specific treatment. We will be coding therapy audio recordings using an adapted TF-CBT Therapy Process Observational Coding System for Children (TF-CBT TPOCS-S) scoring manual. We will also use clinician self-report of fidelity using the Washington State Evidence Based Practice (EBP) Toolkit, and supervisor-report of fidelity in the EBP Toolkit.
  We will ultimately be assessing how fidelity serves as a mediator for the relationship between supervision condition and client outcomes.

SECONDARY OUTCOMES:
Client outcomes for Post-Traumatic Stress and overall functioning | 6 months
  We will complete phone interviews with children and guardians to assess the client outcomes at baseline, 3 months post-baseline, and 6 months post-baseline. We will use the UCLA Post Traumatic Stress Disorder Reaction Index (PTSD RI) to assess trauma exposure and post-traumatic stress symptoms. We will use the Strengths and Difficulties Questionnaire (SDQ), a short behavioral screening survey, to assess overall functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Dorsey, PhD, Principal Investigator — University of Washington; Kelly Thompson, MSW, Study Director — University of Washington
Locations (1):
- University of Washington Department of Psychology, Seattle, Washington, United States

REFERENCES:
- [Derived] Dorsey S, AlRasheed R, Kerns SE, Meza RD, Triplett N, Deblinger E, Jungbluth N, Berliner L, Naithani L, Pullmann MD. A randomized controlled trial testing supervision strategies in community mental health. Implement Res Pract. 2025 May 23;6:26334895251330523. doi: 10.1177/26334895251330523. eCollection 2025 Jan-Dec. PMID 40416801
- [Derived] Dorsey S, Kerns SEU, Lucid L, Pullmann MD, Harrison JP, Berliner L, Thompson K, Deblinger E. Objective coding of content and techniques in workplace-based supervision of an EBT in public mental health. Implement Sci. 2018 Jan 24;13(1):19. doi: 10.1186/s13012-017-0708-3. PMID 29368656
- [Derived] Dorsey S, Pullmann MD, Deblinger E, Berliner L, Kerns SE, Thompson K, Unutzer J, Weisz JR, Garland AF. Improving practice in community-based settings: a randomized trial of supervision - study protocol. Implement Sci. 2013 Aug 10;8:89. doi: 10.1186/1748-5908-8-89. PMID 23937766